CLINICAL TRIAL: NCT04262856
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of AB122 Monotherapy, AB154 in Combination With AB122, and AB154 in Combination With AB122 and AB928 in Front-Line, Non-Small Cell Lung Cancer
Brief Title: Study to Evaluate Monotherapy and Combination Immunotherapies in Participants With PD-L1 Positive Non-small Cell Lung Cancer
Acronym: ARC-7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARC-7 (AB154CSP0002)
Record Dates: First submitted 2020-01-23; First posted 2020-02-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer; Nonsquamous Non Small Cell Lung Cancer; Squamous Non Small Cell Lung Cancer; Lung Cancer
Keywords: Non Small Cell Lung Cancer; Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — zimberelimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (zimberelimab monotherapy) (Experimental): Participants will receive zimberelimab as an intravenous (IV) infusion.
  Interventions: Drug: Zimberelimab
- Arm 2 (domvanalimab and zimberelimab combination therapy) (Experimental): Participants will receive domvanalimab IV in combination with zimberelimab IV infusion.
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- Arm 3 (domvanalimab, etrumadenant, and zimberelimab combination therapy) (Experimental): Participants will receive oral etrumadenant in combination with domvanalimab IV and zimberelimab IV infusion
  Interventions: Drug: Domvanalimab; Drug: Etrumadenant; Drug: Zimberelimab

INTERVENTIONS:
Drug: Domvanalimab — Domvanalimab is a humanized monoclonal antibody targeting human TIGIT
  Other Names: AB154
  Arms: Arm 2 (domvanalimab and zimberelimab combination therapy); Arm 3 (domvanalimab, etrumadenant, and zimberelimab combination therapy)
Drug: Etrumadenant — Etrumadenant is an A2aR and A2bR antagonist
  Other Names: AB928
  Arms: Arm 3 (domvanalimab, etrumadenant, and zimberelimab combination therapy)
Drug: Zimberelimab — Zimberelimab is a fully human anti-PD-1 monoclonal antibody
  Other Names: AB122

SUMMARY:
This randomized phase 2 open-label study will evaluate the safety and efficacy of zimberelimab (AB122) monotherapy, domvanalimab (AB154) in combination with zimberelimab, and domvanalimab in combination with zimberelimab and etrumadenant (AB928) in front-line, PD-L1 positive, metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants; age ≥ 18 years
* Histologically confirmed, treatment naive, metastatic squamous or non-squamous NSCLC with documented high PD-L1 expression, with no epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genomic tumor aberrations.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Must have at least 1 measurable lesion per RECIST v1.1
* Adequate organ and marrow function

Exclusion Criteria:

* Use of any live vaccines against infectious diseases within 28 days of first dose of investigational medicinal products (IMPs)
* Any gastrointestinal condition that would preclude the use of oral medications (eg, difficulty swallowing, nausea, vomiting, or malabsorption)
* History of trauma or major surgery within 28 days prior to the first dose of IMP
* Concurrent medical condition requiring the use of supra-physiologic doses of corticosteroids (> 10 mg/day of oral prednisone or equivalent) or immunosuppressive medications
* Positive test results for Hepatitis B surface antigen, Hepatitis C virus antibody with presence of Hepatitis C qualitative RNA or human immunodeficiency virus (HIV-1 and/or HIV-2) antibody at screening
* Any active autoimmune disease or a documented history of autoimmune disease or syndrome that required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs), except for vitiligo or resolved childhood asthma/atopy.
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From randomization until the first documentation of disease progression or death from any cause, whichever occurs first (up to approximately 3-5 years)
  ORR as assessed by RECIST v1.1
Progression-free survival (PFS) | From randomization until the first documentation of disease progression or death from any cause, whichever occurs first (up to approximately 3-5 years)
  PFS as assessed by RECIST v1.1

SECONDARY OUTCOMES:
Duration of response (DoR) | From the date of first occurrence of a documented objective response to first documentation of disease progression or death from any cause, whichever occurs first (up to approximately 3-5 years)
  DoR as assessed by RECIST v1.1
Disease control rate (DCR) | From the date of first occurrence of a documented objective response to first documentation of disease progression or death from any cause, whichever occurs first (up to approximately 3-5 years)
  DCR as assessed by RECIST v1.1
Overall Survival (OS) | From randomization to death from any cause (up to approximately 5 years)
  OS as assessed at the time of PFS
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | From Screening until up to 90-100 days after the last dose (approximately 5 years)
  The number and percentage of participants that experience TEAE
Pharmacokinetics of zimberelimab | Collected during all treatment cycles (each cycle is 21 or 28 days), up to 14 days post last dose, 30, 60 and 100 days post last dose (in total, an average of 2 years)
  Serum concentration of zimberelimab as determined by validated assays
Pharmacokinetics of domvanalimab | Collected during all treatment cycles (each cycle is 21 or 28 days), up to 14 days post last dose, 30, 60 and 100 days post last dose (in total, an average of 2 years)
  Serum concentration of domvanalimab as determined by validated assays
Pharmacokinetics of etrumadenant | Collected during all treatment cycles (each cycle is 21 or 28 days), up to 14 days post last dose, 30, 60 and 100 days post last dose (in total, an average of 2 years)
  Serum concentration of etrumadenant as determined by validated assays
Immunogenicity of zimberelimab | Collected during all treatment cycles (each cycle is 21 or 28 days), up to 14 days post last dose, 30, and 100 days post last dose (in total, an average of 2 years).
  Percentage of participants who develop treatment-emergent anti-drug antibodies to zimberelimab
Immunogenicity of domvanalimab | Collected during all treatment cycles (each cycle is 21 or 28 days), up to 14 days post last dose, 30, and 100 days post last dose (in total, an average of 2 years).
  Percentage of participants who develop treatment-emergent anti-drug antibodies to domvanalimab

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (44):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Innovative Clinical Research Institute (ICRI), Whittier, California
  - Florida Cancer Specialists, Englewood, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Florida Cancer Specialists - Panhandle, Tallahassee, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - The Valley Hospital - Valley Health System - The Robert and Audrey Luckow Pavilion, Ridgewood, New Jersey
  - Clinical Research Alliance, Lake Success, New York
  - Northwell Health Cancer Institute, Lake Success, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Allegheny General Hospital (AGH)-Alleghney Singer Research Institute, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The Center For Cancer And Blood Disorders (Texas Cancer Care), Fort Worth, Texas
  - Millennium Oncology, Houston, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (4):
  - Border Medical Oncology, Albury
  - Coffs Harbour Health Campus, Coffs Harbour
  - Adelaide Cancer Centre, Elizabeth Vale
  - Shoalhaven Cancer Care Centre, Nowra
- McGill University Health Centre (MUHC) - The Montreal Children's Hospital (MCH), Montreal, Canada
- Hong Kong (2):
  - Hong Kong United Oncology Centre, Hong Kong
  - Queen Elizabeth Hospital (Hong Kong), Hong Kong
- Curie Oncology, Singapore, Singapore
- South Korea (11):
  - Kosin University Gospel Hospital, Busan
  - Chungbuk National University Hospital (CBNUH), Cheongju-si
  - Chonnam University Hospital, Hwasun
  - Gachon University Gil Medical Center, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - St Vincent Hospital of the Catholic University of Korea, Suwon
  - Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
- Taiwan (6):
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Chi Mei Hospital, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-7 - Public website — https://trials.arcusbio.com/study/?id=ARC-7